CLINICAL TRIAL: NCT00092755
Title: A 12-Week, Randomized, Placebo- and Active-Comparator-Controlled, Parallel-Group, Double-Blind Study to Assess the Safety and Efficacy of Etoricoxib 30 mg Versus Ibuprofen 2400 mg in Patients With Osteoarthritis (Study 2)
Brief Title: An Investigational Drug in Patients With Osteoarthritis (0663-073)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0663-073; 2004_056
Record Dates: First submitted 2004-09-23; First posted 2004-09-28 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Osteoarthritis
Keywords: Arcoxia
MeSH Terms: conditions — Osteoarthritis | interventions — Etoricoxib

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0663, etoricoxib
Drug: Comparators: ibuprofen and placebo

SUMMARY:
This study was conducted to assess the safety and tolerability of an investigational drug and to evaluate its effectiveness in the treatment of osteoarthritis of the hip or knee in both men and women.

DETAILED DESCRIPTION:
The duration of treatment is 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with osteoarthritis of the hip or knee who use current approved medication (nonsteroidal anti-inflammatory drugs (NSAIDs)) or tylenol to treat the symptoms of their osteoarthritis. Patients taking NSAIDs are required to discontinue using these drugs and their symptoms must become worse.

Exclusion Criteria:

* Patients with certain medical conditions may not be allowed to participate. These conditions will be reviewed with the study physician.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 548 (Actual)
Dates: Start 2003-04-09 (Actual); Primary Completion 2003-11-13 (Actual); Study Completion 2003-11-13 (Actual)

PRIMARY OUTCOMES:
WOMAC VA 3.0 pain subscale, WOMAC VA 3.0 physical function subscale, and Patient Global Assessment of Disease Status Scale. Efficacy data collected at Weeks 2, 4, 8, and 12.

SECONDARY OUTCOMES:
Patient Global Assessment of Response to Therapy, Investigator Global Assessment of Disease Status, Womac VA 3.0: Stiffness, Overall Average Score and Overall Subscale Average. Clinical efficacy data collected at Weeks 2, 4, 8, and 12.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Puopolo A, Boice JA, Fidelholtz JL, Littlejohn TW, Miranda P, Berrocal A, Ko A, Cichanowitz N, Reicin AS. A randomized placebo-controlled trial comparing the efficacy of etoricoxib 30 mg and ibuprofen 2400 mg for the treatment of patients with osteoarthritis. Osteoarthritis Cartilage. 2007 Dec;15(12):1348-56. doi: 10.1016/j.joca.2007.05.022. Epub 2007 Jul 16. PMID 17631392